CLINICAL TRIAL: NCT01094275
Title: Role of CYP2C19 Polymorphism in the Drug Interaction Between Clopidogrel and Omeprazole
Status: Completed | Type: Observational
Sponsor: Neil Kleiman, MD (Other)
Responsible Party: Sponsor-Investigator, Neil Kleiman, MD, Professor of Medicine Weill Cornell Medical College Medical Director Cardiac Catheterization Laboratories, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00003846
Record Dates: First submitted 2010-02-10; First posted 2010-03-26 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
Keywords: drug resistance; gene polymorphism
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Omeprazole

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: None Retained — Cheek swabs for DNA, blood samples for drug metabolite estimation and platelet function study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- wild / normal type allele of CYP2C gene: clopidogrel 75 mg alone.
  Interventions: Drug: Clopidogrel 75mg, Omeprazole 20mg
- wild / normal type allele of CYP2C: clopidogrel 75 mg + omeprazole 20 mg.
  Interventions: Drug: Clopidogrel 75mg, Omeprazole 20mg
- Loss of Haplotype CYP2C19: clopidogrel 75mg alone
  Interventions: Drug: Clopidogrel 75mg, Omeprazole 20mg
- Loss of function haplotype of CYP2C: clopidogrel 75mg + omerprazole 20mg.
  Interventions: Drug: Clopidogrel 75mg, Omeprazole 20mg

INTERVENTIONS:
Drug: Clopidogrel 75mg, Omeprazole 20mg — Clopidogrel and or Omeprazole as applicable
  Other Names: Plavix , Prilosec OTC

SUMMARY:
Clopidogrel, an inhibitor of ADP induced platelet aggregation and activation, is one of the most commonly used drugs in patients with cardiovascular disease. The specific aim of the proposed study is to determine whether the interaction between proton-pump inhibitors (PPIs) and clopidogrel is dependent on CYP2C19 haplotype.

DETAILED DESCRIPTION:
Clopidogrel, an inhibitor of ADP induced platelet aggregation and activation, is one of the most commonly used drugs in patients with cardiovascular disease; coronary-stenting would not be possible without the robust anti platelet function of this drug. Clopidogrel is a pro-drug that is transformed through a series of hepatic cytochrome p-450 (CYP) enzymes to an active metabolite. One of these CYP enzymes, 2C19 is subject to competitive inhibition by commonly used proton-pump inhibitors (PPIs). PPIs are commonly used for gastro-esophageal protection in patients treated with clopidogrel. Around 63% of 3,799 patients on clopidogrel received a PPI at TMH in 2008.

Recently, a series of publications indicated that clopidogrel active metabolite levels and platelet inhibition are lower in patients receiving PPIs. In addition, a recent survey of >16,690 patients in Medco database indicates that use of PPIs is associated with a 51% increase in the risk of death or myocardial infarction in patients receiving clopidogrel. Recent data have also indicated that patients with loss of function (LOF) haplotypes of the CYP2C19 gene have lower levels of the active metabolite after dosing with clopidogrel. These patients have higher rates of death, myocardial infarction, stent thrombosis and other ischemic complications than do patients with the wild type enzyme. Inadequate responses to clopidogrel therapy have been implicated as an important predictor of adverse clinical events. The reported prevalence of non-responsiveness to clopidogrel among patients with cardiovascular disease is between 4% and 34%, depending on the method and definition used to assess this parameter. Approximately 25% of American population carries a LOF mutation of CYP2C19.

It is unclear whether the concomitant use of omeprazole (PPI) with clopidogrel would result in a decrease in platelet function parameters through the CYP2C19 clopidogrel activation pathway. The specific aim of the proposed study is to determine whether the interaction between PPIs and clopidogrel is dependent on CYP2C19 haplotype. We hypothesize that among subjects with a LOF genotype, the interaction between clopidogrel and PPIs is greater than that in subjects with the wild type genotype7 and is manifest in both platelet function parameters and in conversion of clopidogrel to its active metabolite.

Approximately 75 randomly selected healthy volunteer subjects will be screened with the intent of identifying at least 16 subjects who are heterozygous for a LOF mutation of CYP2C19 (known as *2/rs4244285, *3).

Subjects with the LOF allele will be selected along with age and gender-matched wild type controls and baseline platelet function studies will be performed (n=16 for each group). Subjects in each stratum will then be randomly assigned to receive one week of clopidogrel in combination with omeprazole or clopidogrel alone. Subjects initially assigned to clopidogrel + omeprazole will then take clopidogrel only and subjects initially assigned to clopidogrel only will take both clopidogrel and omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* age 18- 65
* healthy - not taking any drugs / over the counter drugs regularly.
* ability and commitment to take the drugs and volunteer for 3 blood draws.

Exclusion Criteria:

* Taking any scheduled medication known to affect platelet function such as clopidogrel or NSAIDS11, COX2 inhibitors, beta blockers, calcium channel blockers, diuretics, anti-coagulants, older psychotropic agents, and recent ingestion of alcohol and caffeine
* Known history of heart disease
* Bleeding disorders
* Known allergy or contraindications to omeprazole or clopidogrel
* Pregnant and nursing women will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects aged 18-65.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
The effect of omeprazole on platelet inhibition by clopidogrel | 3 weeks
  To test whether concomitant administration of omeprazole will decrease the platelet inhibitory properties of clopidogrel in subjects with LOF mutation of CYP2C19 (known as *2 and *3)

SECONDARY OUTCOMES:
The effect of omeprazole on the conversion of clopidogrel | 3 weeks
  To test whether concomitant administration of omeprazole will decrease the conversion of clopidogrel to its active metabolite in subjects with loss of function (LOF) mutation of CYP2C19 (known as *2 and *3)

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Kleiman, MD, Principal Investigator — Methodist DeBakey Heart Center.
Locations (1):
- The Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data to be determined.

REFERENCES:
- [Background] Srinivas Nadipalli, Sashidar Guthikonda, Timothy R. DelaO, Ali J. Marian, Federico Monzon, Ping Wang, Neal S. KleimanDOES A LOSS OF FUNCTION POLYMORPHISM OF CYP2C19 MODULATE THE EFFECTS OF CLOPIDOGREL. J Am Coll Cardiol. 2011;57 E1201.